CLINICAL TRIAL: NCT05186389
Title: Jejunal Luminal and Colonic Mucosa-Associated Microbiota in Metabolic Diseases: Methods, Identification and Causalities
Acronym: JE/COL-MIME
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-86
Record Dates: First submitted 2021-12-07; First posted 2022-01-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus; Obesity; Metabolic Disease
Keywords: microbiota; endoscopy; colonoscopy; obesity; type II diabetes
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Metabolic Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Saliva, urines, blood, jejunal fluid, jejunal biopsies, colonic biopsies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- "Control Group": 15 non-obese participants considered "metabolically-healthy" : "control group"
- Obese group (Ob): 15 severely obese participants, candidates for bariatric surgery, but without T2D: "obese group" (Ob)
- Obese and Type 2 Diabetes group (ObD): 15 participants who are both severely obese, candidates for bariatric surgergy and diagnosed with T2D: "obese and diabetic group" (ObD).

SUMMARY:
This clinical study will investigate Jejunal Microbiota in Metabolic Diseases (Je-MiMe, n=45) and Colonic mucosa-associated Microbiota in Metabolic Diseases (Col-MiMe, n=45).

Each cohort (Je and Col -MiMe) is composed of three groups: participants with obesity (n=15) with obesity and with type II diabetes (n=15).

This research protocol is organized in two parts. Each part of this study will recruit 45 participants that are only recruited in one of the parts of the protocol (JE-MIME or COL-MIME). Thus, in total, the study will include 90 patients. Each part of this study is composed of 3 groups: 1) "Control Group ", 2) Obese group (Ob), 3) Obese and Type 2 Diabetes group (ObD). Control groups for part I (JE-MIME) and part 2 (COL-MIME) are composed of different participants. Each group is composed of 15 human adult volunteers for the JE-MIME study (part 1) and 15 participants for the COL-MIME study (part 2). Total number of participants is 45 for part 1, and 45 for part 2. Total number for this project is 90.

Microbiota wil be collected during an endoscopy or coloscopy which is planned as routine care for the patients.

Primary objectives are to characterize jejunal (JE-MIME, Part I of the study) and colonic mucosa-associated microbiota (COLMIME, Part II of the study) and compare both microbiota to faecal microbiota (evaluate differences and similarities between jejunal microbiota or mucus-associated microbiota and faecal microbiota).

Secondary objectives are to 1) Correlate microbiota with metabolic health and inflammatory markers; 2) Correlate microbiota with lifestyle and neuropsychological health.

Both the jejunal microbiota and mucus-associated microbiota are strong integrators of nutritional environment and intestinal health status, respectively, compared to the fecal microbiota. This study will help to better understand the physiopathology of metabolic diseases. This research could lead to finding specific microbiota members, either from the jejunal compartment or from the inner mucus layer, crucial for the promotion / protection of chronic intestinal inflammation and associated metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

  * Aged between 18 and 60 years;
  * Ability to understand and provide informed consent (in French);
  * Ability and willingness to meet the required schedule and study procedures;
* Group-Specific Inclusion Criteria:
* Control Group

Inclusion criteria for the participants from the Control group are:

* Presence of Gastroesophageal Reflux Disease symptoms or gastric discomfort.
* BMI [19kg/m² < BMI <25 kg/m²]
* Match age and sex to the patients from the Ob and ObD groups.
* Only patients with normal glucose tolerance (NGT), glucose tolerance (IGT) and/or fasting glucose (IFG) and an HbA1c < 6.5 % will be included in this group.

  * Ob Group

Inclusion criteria for the participants from Ob and ObD groups are:

● Candidate for bariatric surgery and meet the HAS criteria (Haute Autorité de Santé, 2009) :

* IMC ≥ 40 kg/m² without comorbidities Or IMC≥ 35 kg/m² with at least one obesity-related comorbidity (i.e.: Hypertension, Dyslipidemia, Obstructive Sleep Apnea, Joints Disease, non-alcoholic steatohepatitis, excluding T2D)
* Weight stable for at least 2 months
* No treatment for metabolic health complications, no previous obesity surgery, no obesity treatment drug.
* No monogenic form of obesity (Hebebrand et al., 2017)

  * ObD Group

Inclusion criteria for the participants from ObD groups are:

* Candidate for bariatric surgery with T2D
* At least one obesity-related comorbidity including T2D
* Fasting plasma glucose (FPG) ≥7 mM (=1.26g/l) or
* Participants with HbA1c ≥ 6.5% (48 mmol/mol)
* All stages of albuminuria

Exclusion Criteria:

* General Non-inclusion Criteria:

  * Treatment for the previous 12 week that could

    * alter gastrointestinal motor function (e.g. opioids, prokinetics, anticholinergics, laxatives),
    * acidity (PPI, H2RA)
    * microbial population (e.g.: antibiotics, probiotics)
    * immunosuppressants (eg: calcineurin inhibitors, corticosteroids, biological agents, etc.).
    * use of weight-loss drug or dietary intervention aiming to lose weight;
  * Altered anatomy of the esophagus, stomach, small or large intestine due to prior gastrointestinal surgery (exceptions include appendectomy or cholecystectomy more than 3 months prior to enrollment) or other reasons;

    * Any abdominal or pelvic surgery within the past 3 months;
    * Diverticulitis, diverticular stricture, or other intestinal strictures.
    * Intestinal resection of the gastrointestinal tract
  * Previous history of gastric bezoar or gastroparesis
  * Acute or chronic inflammatory bowel disease or infections diseases (i.e.: VHC, VHB, VIH, etc.)
  * Abdominal or pelvic radiotherapy or abdominal cancer
  * Colorectal cancer, either known or not
  * Dysphagia, eosinophilic esophagitis, esophageal stricture, or other swallowing disorder
  * Organ Transplantation and patients on Immunosuppressive Therapy
  * Severe kidney failure and/or patients on dialysis therapy (serum creatinine > 150 μmol/l or eGFR < 60 ml/min per 1.73 m2 body surface area)
  * CVD, endocrine, renal or other chronic disease likely to affect motility.
  * Colon cleansing preparation during the last 1 month
  * No < 3 bowel movements per week
  * Females of childbearing age who do not practice birth control and/or are pregnant or lactating
  * Participants non-affiliated to the French national health scheme
  * Participants who are already included in a clinical study which implies testing any pharmaceutical drug.
  * Participants who do not understand the research procedures those who are institutionalized, or who unable to give informed consent
  * Participants placed under legal protection
  * Patients with drug addiction
  * Antibiotherapy 3 months preceding the endoscopy
  * Weight variation (diminution or increase) > 5kg in the last 3 months
* Specific non-inclusion Criteria
* Ob and ObT2D Group

  * Usual contraindication for bariatric surgery;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Control Group 15 non-obese participants considered "metabolically-healthy" : "control group"
  2. Obese group (Ob) 15 severely obese participants, candidates for bariatric surgery, but without T2D: "obese group" (Ob)
  3. Obese and Type 2 Diabetes group (ObD) 15 participants who are both severely obese, candidates for bariatric surgergy and diagnosed with T2D: "obese and diabetic group" (ObD).
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Metagenomic analysis | 1 month
  Single time point analysis of jejunal or colonic mucosal-associated and fecal microbiota.
  Microbiota will be analysed through 16S rRNA gene sequencing as well as shotgun metagenomic sequencing of the different samples.
  We will examine if jejunal microbiota abundance is decreased in subjects with obesity and obesity + type 2 diabetics compared to lean subjects. Based on metagenomic sequencing data, the number of bacterial genes will be estimated and compared between groups.
  We will examine the distance of bacterial layer in the mucus from intestinal epithelial cells in people with T2D as compared to people without T2D and lean subjects.

SECONDARY OUTCOMES:
Clinical associations with metagenomic analysis | 1 month
  Single time point analysis : Investigation of the correlations between jejunal microbiota or mucosal-associated microbiota and clinical parameters.
  Secondary objectives are to analyse the relationship between jejunal microbiota/mucus-associated microbiota and metabolic health, inflammation, lifestyle and mental health that will be evaluated through extensive bio-clinical phenotyping and will include:
  * Metabolic phenotype (serum)
  * Systemic inflammation status and Entero and Neuroendocrine markers (serum and biopsies)
  * Anthropometric measurements
  * Histological analysis of the jejunal biopsy obtained during endoscopy and colonoscopy
  * Lifestyle factors collected through lifestyle questionnaires:
    * Medical history questionnaires
    * Dietary patterns
    * Physical activity
    * Smoking habits
    * Psycho-emotional health and Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé des Peupliers, 8 Place de l'Abbé Georges Hénocque, 75013, Paris, France